CLINICAL TRIAL: NCT02883309
Title: Efficacy of an Intradialysis Combined Muscle Strength and Cardiorespiratory Capacity Training Program on Disability Level and Physical Performance, in Patients With Chronic Renal Failure at a Kidney Replacement Therapy Unit.
Brief Title: Efficacy of an Intradialysis Combined Training Program on Disability Level and Physical Performance.
Acronym: PTH-CKD0113
Status: Approved for marketing | Type: Expanded Access
Sponsor: Universidad Austral de Chile (Other)
Collaborators: Nephrocare Portugal (Industry)
Responsible Party: Sponsor
Other Study IDs: Universidad Austral de Chile; 33-2013 (Other Grant/Funding Number: DE-UACh)
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Renal Failure
Keywords: Hemodialysis; Skeletal muscle; Exercise; Rehabilitation; Disability Evaluation
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity

INTERVENTIONS:
Other: intradialytic physical training program — Nine patients participated in the experimental group in a combined training program, which lasted 12 weeks with a frequency of 3 times a week, the training sessions were carried out within each dialysis session during the first 2 hours of the dialysis treatment, the working session involved a warm up period, aerobic exercise with pedals, or strength exercises based on free weight depending on the training stage. The Borg scale and the heart rate reserve were used to control the training intensity. The disability level was evaluated at the beginning and the end of the study through the World Health Organization Disability Assessment Schedule II, the aerobic capacity was evaluated through the six minute walk and the limbs strength was evaluated through a dynamometer.

SUMMARY:
The patient subjected to hemodialysis has a low physical capacity due to being advanced in years and the complexity of the process, which is encouraged by family members and caregivers who lead them to a total dependence. The Intradialytic physical exercise is presented as an alternative to counteract this functional deterioration of patients with terminal chronic kidney failure.

DETAILED DESCRIPTION:
Objective To evaluate the impact of the intradialytic physical training program on the level of disability and physical performance in patients subjected to hemodialysis.

Materials and methods 18 patients subjected to hemodialysis, whose ages ranged from 54 to 84 (10 women) were included in the study. Nine of these patients participated in a combined training program, which lasted 12 weeks, the training sessions were carried out within each dialysis session, the working session involved a warm-up period, aerobic exercise with pedals, or strength exercises based on free-weight depending on the training stage. The Borg scale and the heart rate reserve were used to control the training intensity. The disability level was evaluated at the beginning and end of the study through the World Health Organization Disability Assessment Schedule II, the six minutes walk test (6MWT), quadriceps strength, Kt/V, serum levels of potassium and creatinine.

Outcomes One subject belonging to the experimental group did not complete the training due to problems in the venous access during the 1st month of training. 8 patients in to the experimental group showed significant improvements in the 6MWT, quadriceps strength and decrease in the level of disability. No changes were observed in the control group. No significant changes were found in the serum levels of potassium and creatine.

Conclusions An Intradialytic physical training program achieved a substantial decrease in the level of disability, and an improvement of aerobic capacity and muscle strength. The study was funded by the extension office of the Austral University of Chile.

ELIGIBILITY:
Inclusion Criteria:

* Patients which are subject to process of hemodialysis via arteriovenous fistula in dialysis unit Valdivia.
* Which are between 60-80 years.
* Therapy Dialysis for more than 3 months period.
* Submit 24 or more points on the Mini-mental state test.

Exclusion Criteria:

* Inability to understand orders.
* Dyspnea at rest.
* Hospitalized one month before surgery.
* Diseases Cerebrovascular transient ischemic attacks.
* Lower limb amputation (ankle presence) that this orthopedic prosthesis.
* Syndrome Acute coronary.
* Congestive heart failure or severe pneumonia.
* Patients with uncontrolled diabetes pharmacologically or are not within the appropriate standards of glucose for training.
* Patients with uncontrolled hypertension pharmacologically or are not within the proper blood pressure standards for training.
* Persistent Hyperkalemia .
* Angina at rest.
* Lung-disease which results in adverse effects.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula I Moscoso, Mph PTh, Study Chair — Universidad Austral de Chile; Roberto G Mancilla, Student, Principal Investigator — Universidad Austral de Chile; Cesar E Gonzalez, Student, Principal Investigator — Universidad Austral de Chile; Manuel Monrroy, Msc(c) PTh, Study Director — Universidad Austral de Chile; Lizzy Orellana, MD, Study Director — Universidad Austral de Chile

REFERENCES:
- [Background] Marriott HE, Lamb KL. The use of ratings of perceived exertion for regulating exercise levels in rowing ergometry. Eur J Appl Physiol Occup Physiol. 1996;72(3):267-71. doi: 10.1007/BF00838650. PMID 8820897
- [Background] Johansen KL, Shubert T, Doyle J, Soher B, Sakkas GK, Kent-Braun JA. Muscle atrophy in patients receiving hemodialysis: effects on muscle strength, muscle quality, and physical function. Kidney Int. 2003 Jan;63(1):291-7. doi: 10.1046/j.1523-1755.2003.00704.x. PMID 12472795
- [Background] Kurella Tamura M, Covinsky KE, Chertow GM, Yaffe K, Landefeld CS, McCulloch CE. Functional status of elderly adults before and after initiation of dialysis. N Engl J Med. 2009 Oct 15;361(16):1539-47. doi: 10.1056/NEJMoa0904655. PMID 19828531
- [Background] Johansen KL. Physical functioning and exercise capacity in patients on dialysis. Adv Ren Replace Ther. 1999 Apr;6(2):141-8. doi: 10.1016/s1073-4449(99)70032-4. PMID 10230881
- [Background] de Lima MC, Cicotoste Cde L, Cardoso Kda S, Forgiarini LA Jr, Monteiro MB, Dias AS. Effect of exercise performed during hemodialysis: strength versus aerobic. Ren Fail. 2013;35(5):697-704. doi: 10.3109/0886022X.2013.780977. Epub 2013 Apr 8. PMID 23560491
- [Background] Ribeiro R, Coutinho GL, Iuras A, Barbosa AM, Souza JA, Diniz DP, Schor N. Effect of resistance exercise intradialytic in renal patients chronic in hemodialysis. J Bras Nefrol. 2013 Jan-Mar;35(1):13-9. doi: 10.5935/01012800.20130003. English, Portuguese. PMID 23598747
- [Background] Giannaki CD, Stefanidis I, Karatzaferi C, Liakos N, Roka V, Ntente I, Sakkas GK. The effect of prolonged intradialytic exercise in hemodialysis efficiency indices. ASAIO J. 2011 May-Jun;57(3):213-8. doi: 10.1097/MAT.0b013e318215dc9e. PMID 21412149
- [Background] KARVONEN MJ, KENTALA E, MUSTALA O. The effects of training on heart rate; a longitudinal study. Ann Med Exp Biol Fenn. 1957;35(3):307-15. No abstract available. PMID 13470504
- [Background] American College of Sports Medicine Position Stand. The recommended quantity and quality of exercise for developing and maintaining cardiorespiratory and muscular fitness, and flexibility in healthy adults. Med Sci Sports Exerc. 1998 Jun;30(6):975-91. doi: 10.1097/00005768-199806000-00032. PMID 9624661
- [Background] Stoudemire NM, Wideman L, Pass KA, McGinnes CL, Gaesser GA, Weltman A. The validity of regulating blood lactate concentration during running by ratings of perceived exertion. Med Sci Sports Exerc. 1996 Apr;28(4):490-5. doi: 10.1097/00005768-199604000-00014. PMID 8778555
- [Background] Mercer TH, Naish PF, Gleeson NP, Wilcock JE, Crawford C. Development of a walking test for the assessment of functional capacity in non-anaemic maintenance dialysis patients. Nephrol Dial Transplant. 1998 Aug;13(8):2023-6. doi: 10.1093/ndt/13.8.2023. PMID 9719158
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] DePaul V, Moreland J, Eager T, Clase CM. The effectiveness of aerobic and muscle strength training in patients receiving hemodialysis and EPO: a randomized controlled trial. Am J Kidney Dis. 2002 Dec;40(6):1219-29. doi: 10.1053/ajkd.2002.36887. PMID 12460041
- [Background] Headley S, Germain M, Mailloux P, Mulhern J, Ashworth B, Burris J, Brewer B, Nindl BC, Coughlin M, Welles R, Jones M. Resistance training improves strength and functional measures in patients with end-stage renal disease. Am J Kidney Dis. 2002 Aug;40(2):355-64. doi: 10.1053/ajkd.2002.34520. PMID 12148109
- [Background] Parsons TL, Toffelmire EB, King-VanVlack CE. Exercise training during hemodialysis improves dialysis efficacy and physical performance. Arch Phys Med Rehabil. 2006 May;87(5):680-7. doi: 10.1016/j.apmr.2005.12.044. PMID 16635631
- [Background] Redelmeier DA, Bayoumi AM, Goldstein RS, Guyatt GH. Interpreting small differences in functional status: the Six Minute Walk test in chronic lung disease patients. Am J Respir Crit Care Med. 1997 Apr;155(4):1278-82. doi: 10.1164/ajrccm.155.4.9105067.
- [Background] Posl M, Cieza A, Stucki G. Psychometric properties of the WHODASII in rehabilitation patients. Qual Life Res. 2007 Nov;16(9):1521-31. doi: 10.1007/s11136-007-9259-4. Epub 2007 Sep 9. PMID 17828578
- [Background] Garin O, Ayuso-Mateos JL, Almansa J, Nieto M, Chatterji S, Vilagut G, Alonso J, Cieza A, Svetskova O, Burger H, Racca V, Francescutti C, Vieta E, Kostanjsek N, Raggi A, Leonardi M, Ferrer M; MHADIE consortium. Validation of the "World Health Organization Disability Assessment Schedule, WHODAS-2" in patients with chronic diseases. Health Qual Life Outcomes. 2010 May 19;8:51. doi: 10.1186/1477-7525-8-51. PMID 20482853
- See also: Estudio piloto sobre entrenamiento físico durante hemodiálisis — http://www.scielo.cl/scielo.php?pid=S0034-98872011000800010&script=sci_arttext
- See also: Whodas II Acta Psiquiatrica — https://www.google.cl/url?sa=t&rct=j&q=&esrc=s&source=web&cd=1&cad=rja&uact=8&ved=0CB4QFjAA&url=http%3A%2F%2Fwww.researchgate.net%2Fprofile%2FLuis_Gaite%2Fpublication%2F230554738_Version_en_lengua_espaola_de_un_nuevo_cuestionario_de_evaluacion_de_disca
- See also: Intradialytic versus home based exercise training in hemodialysis patients: a randomised controlled trial — http://www.biomedcentral.com/1471-2369/10/2
- See also: Efeitos do exercício físico durante a hemodiálise em indivíduos com insuficiência renal crônica: uma revisão — http://www.revistas.usp.br/fpusp/article/view/12081